CLINICAL TRIAL: NCT02661581
Title: Peer-led, Empowerment-based, Approach to Self-management Efforts in Diabetes: A Pragmatic Trial
Brief Title: Peer-led, Empowerment-based, Approach to Self-management Efforts in Diabetes
Acronym: PLEASED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: VGH and UBC Hospital Foundation (Other)
Responsible Party: Principal Investigator, Tricia Tang, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H13-02163-A002
Record Dates: First submitted 2015-02-24; First posted 2016-01-22 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Diabetes
Keywords: Diabetes; Peer Leader Support
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Support (Experimental): Peer support intervention group: During the first 3 months of DSME, participants in the DSMS intervention group will be invited to attend 6 lifestyle change sessions delivered a 2-person peer leader team and conducted bi-weekly. Immediately following the 3 months of DSME, participants are invited to attend 9 months of weekly DSMS sessions (60-minutes per session) delivered by a Peer Leader. These sessions are designed to sustain the self-management gains achieved in the 3 months of DSME.
  Interventions: Behavioral: Peer Support
- Control (No Intervention): Immediately following the 6 bi-weekly DSME sessions, participants randomized to the control group will have completed their participation in the study.

INTERVENTIONS:
Behavioral: Peer Support — The intervention is lifestyle change. First, the peer leaders will be trained how to conduct diabetes self-management education and support sessions. During the first 3 months, all the participants will attend the diabetes self-management education sessions. The participants in the intervention arm will also receive diabetes self-management support sessions as well. In the end of the first 3 months, the intervention group participants will receive weekly support sessions for 9 months.
  Arms: Peer Support

SUMMARY:
PLEASED is a 12-month program that aims to help South Asians with type 2 diabetes improve and sustain diabetes-related health outcomes e.g. glycemic control, quality of life...) achieved from previous short-term diabetes education program. Our goal is to provide a new generation of education and support that can be ongoing, patient-driven, and flexible to the dynamic and evolving conditions of patients' "real-word" environment and life circumstances.

DETAILED DESCRIPTION:
Diabetes self-management education: In the first three months of PLEASED, patients with type 2 diabetes will participate in 12 weekly sessions: 6 sessions will focus on diabetes education and be delivered by a health professional and 6 sessions will focus on lifestyle change and be delivered by a peer leader. Education sessions will be 2-hours long and be facilitated by nurses, dieticians, and pharmacists. Patients will learn about the diabetes disease process, lifestyle modification, healthy eating, physical activity, medications, monitoring, short- and long- complications, diabetes distress, and coping. Lifestyle change sessions will be 1-hour long and start with 30 minutes of physical activity followed by 30 minutes of goal-setting, action planning, and problem solving. Additional activities such as recipe makeovers and exchanges will also be included.

Diabetes self-management support: In the next nine months of the PLEASED program, patients will be invited to attend 32 weekly self-management support sessions (1-hour long) facilitated by a peer leader. The goal of these sessions is to help patients continue making positive lifestyle changes. Each support session will start with 30 minutes of physical activity led by the peer leader followed by a discussion where participants are invited to (1) discuss self-management challenges, (2) share thoughts and feelings about these challenges, (3) ask self-management questions, (4) engage in problem solving, and (5) set self-management goals and design behavioral experiments to achieve those goals. Patients are invited to attend as frequently as they need or as they are able to given other competing life demands. While these sessions focus on lifestyle change and emotional support, participants will be able to obtain responses to medical and clinical questions from 811 or the PLEASED hotline (hosted by dieticians, nurses, and pharmacists).

All patients enrolled in the PLEASED program will undergo three free health assessments: at the start of the program, at 3 months, and at 12 months. Health assessments will include measuring glycemic control, ApoB, blood pressure, waist circumference, weight, and body mass index. All patients will also complete a survey assessing quality of life, social support, depression, and self-efficacy.

ELIGIBILITY:
To be eligible to participate as a subject in this study, individuals must

1. Have type 2 diabetes,
2. Be of South Asian background,
3. Live in the Metro Vancouver area,
4. Be at least 21 years old,
5. Have transportation to attend group sessions.

To be eligible to participate as a peer leader in this study, individuals must

1. Have diabetes or are a caregiver to someone who has diabetes,
2. Are of South Asian background,
3. Live in the Greater Vancouver area,
4. Are at least 21 years old,
5. Are bilingual in English and Punjabi,
6. Have transportation to attend training,
7. Are able and willing to commit to 6 sessions of training (5 hours each, over a 6 week period)

Exclusion criteria for both participants and peer leaders include:

1. Serious health conditions
2. Addictions to alcohol or drugs, which would hinder meaningful participation in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Glycemic Control measured by HbA1c | Up to 12 months
  To compare a peer support model for diabetes self-management support (DSMS) to usual care on sustaining improvements in glycemic control achieved from short-term diabetes self-management education (DSME).

SECONDARY OUTCOMES:
Blood pressure (mmHg) measured by Omron BP785 monitor | Up to 12 months
ApoB (g/L) will be collected using venous puncture blood draw | Up to 12 months
Waist circumference (inch) measured by Seca 203 Circumference Measuring Tape | Up to 12 months
Body Mass Index (kg/m2) | Up to 12 months
Physical activity measured by the actical accelerometer | Up to 12 months
Diabetes-specific Social Support will be assessed using a 4-item perceived social support scale developed by Tang et al. that measures amount of support and satisfaction with support from family, friends and the health care team | Up to 12 months
Depressive Symptom Severity will be assessed with the PRIME-MD Patient Health Questionnaire (PHQ-9) | Up to 12 months
Diabetes-related distress measured by the Diabetes Distress Scale (DDS), a 17-item scale developed by Polonsky and colleagues | Up to 12 months
Height measured using a stadiometer | Up to 12 months
Weight measured on a high quality, calibrated digital scale, with the participant wearing clothes, but no shoes | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Tang, PhD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada